CLINICAL TRIAL: NCT02388061
Title: Extending the Time for Thrombolysis in Emergency Neurological Deficits - Intra-Arterial Using Intravenous Tenecteplase
Brief Title: Tenecteplase Versus Alteplase Before Endovascular Therapy for Ischemic Stroke
Acronym: EXTEND-IA TNK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuroscience Trials Australia (Other)
Collaborators: The Florey Institute of Neuroscience and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTA1401
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous tenecteplase (TNK) (Experimental): Patients will receive intravenous tenecteplase (0.25mg/kg, maximum 25mg, administered as a bolus over ~10 seconds).
  Interventions: Drug: Tenecteplase
- Intravenous tissue plasminogen activator (tPA) (Active Comparator): Patients will receive intravenous t-PA at the standard licensed dose of 0.9 mg/kg up to a maximum of 90mg, 10% as bolus and the remainder over 1 hour.
  Interventions: Drug: Tissue Plasminogen Activator

INTERVENTIONS:
Drug: Tenecteplase
  Other Names: TNK
  Arms: Intravenous tenecteplase (TNK)
Drug: Tissue Plasminogen Activator
  Other Names: Alteplase; tPA
  Arms: Intravenous tissue plasminogen activator (tPA)

SUMMARY:
Patients presenting to the emergency department with acute ischemic stroke, who are are eligible for standard intravenous tPA therapy within 4.5 hours of stroke onset will be assessed for major vessel occlusion to determine their eligibility for randomization into the trial. If the patient gives informed consent they will be randomised 50:50 using central computerised allocation to intravenous alteplase or tenecteplase before all participants undergo intra-arterial clot retrieval. The trial is prospective, randomised, open-label, blinded endpoint (PROBE) design.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with acute ischemic stroke eligible using standard criteria to receive IV thrombolysis within 4.5 hours of stroke onset
2. Patient's age is ≥18 years
3. Intra-arterial clot retrieval treatment can commence (arterial puncture) within 6 hours of stroke onset.
4. Arterial occlusion on CTA or MRA of the ICA, M1, M2 or basilar artery.

Exclusion Criteria:

1. Intracranial hemorrhage (ICH) identified by CT or MRI
2. Rapidly improving symptoms at the discretion of the investigator
3. Pre-stroke mRS score of ≥ 4 (indicating previous disability)
4. Hypodensity in >1/3 MCA territory or equivalent proportion of basilar artery territory on non-contrast CT
5. Contra indication to imaging with contrast agents
6. Any terminal illness such that patient would not be expected to survive more than 1 year
7. Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.
8. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with substantial angiographic reperfusion (mTICI) score of 2b/3 (restoration of blood flow to >50% of the affected arterial territory) or absence of retrievable thrombus at initial angiogram. | Initial angiogram (day 0)

SECONDARY OUTCOMES:
Proportion of patients with ≥8 point reduction in NIHSS or reaching 0-1 at 3 days (favourable clinical response) adjusted for baseline NIHSS and age. | Initial angiogram (day 0)
Modified Rankin Scale (mRS) at 3 months | 3 months post stroke
  ordinal analysis
mRS 0-1 or no change from baseline at 3 months | 3 months post stroke
mRS 0-2 or no change from baseline at 3 months | 3 months post stroke
Symptomatic intracranial hemorrhage (SICH) | within 36 hours post treatment
Death due to any cause | Up to 3 months post stroke
Proportion of patients with angiographic reperfusion adjusted for hyperdense clot length on non-contrast CT and time from thrombolysis to initial angiogram | Up to 24 hours post treatment

CONTACTS AND LOCATIONS:
Locations (18):
- Australia (16):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane & Women's Hospital, Brisbane, Queensland
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Western Heath, St Albans, Victoria
- New Zealand (2):
  - Auckland Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch

REFERENCES:
- [Derived] Yogendrakumar V, Beharry J, Churilov L, Pesavento L, Alidin K, Ugalde M, Weir L, Mitchell PJ, Kleinig TJ, Yassi N, Thijs VN, Wu TY, Brown H, Dewey HM, Wijeratne T, Yan B, Sharma GJ, Desmond P, Parsons MW, Donnan GA, Davis SM, Campbell BCV; EXTEND-IA TNK and Royal Melbourne Stroke Registry Investigators. Association of Time to Thrombolysis With Early Reperfusion After Alteplase and Tenecteplase in Patients With Large Vessel Occlusion. Neurology. 2024 Apr 9;102(7):e209166. doi: 10.1212/WNL.0000000000209166. Epub 2024 Mar 19. PMID 38502892
- [Derived] Yogendrakumar V, Churilov L, Mitchell PJ, Kleinig TJ, Yassi N, Thijs V, Wu T, Shah D, Bailey P, Dewey HM, Choi PMC, Ma A, Wijeratne T, Garcia-Esperon C, Cloud G, Chandra RV, Cordato DJ, Yan B, Sharma G, Desmond PM, Parsons MW, Donnan GA, Davis SM, Campbell BCV; EXTEND-IA TNK Investigators. Safety and Efficacy of Tenecteplase and Alteplase in Patients With Tandem Lesion Stroke: A Post Hoc Analysis of the EXTEND-IA TNK Trials. Neurology. 2023 May 2;100(18):e1900-e1911. doi: 10.1212/WNL.0000000000207138. Epub 2023 Mar 6. PMID 36878701
- [Derived] Sarraj A, Albers GW, Mitchell PJ, Hassan AE, Abraham MG, Blackburn S, Sharma G, Yassi N, Kleinig TJ, Shah DG, Wu TY, Hussain MS, Tekle WG, Gutierrez SO, Aghaebrahim AN, Haussen DC, Toth G, Pujara D, Budzik RF, Hicks W, Vora N, Edgell RC, Slavin S, Lechtenberg CG, Maali L, Qureshi A, Rosterman L, Abdulrazzak MA, AlMaghrabi T, Shaker F, Mir O, Arora A, Martin-Schild S, Sitton CW, Churilov L, Gupta R, Lansberg MG, Nogueira RG, Grotta JC, Donnan GA, Davis SM, Campbell BCV; SELECT, EXTEND-IA, EXTEND-IA TNK, and EXTEND-IA TNK Part-II Investigators. Thrombectomy Outcomes With General vs Nongeneral Anesthesia: A Pooled Patient-Level Analysis From the EXTEND-IA Trials and SELECT Study. Neurology. 2023 Jan 17;100(3):e336-e347. doi: 10.1212/WNL.0000000000201384. Epub 2022 Oct 26. PMID 36289001
- [Derived] Yogendrakumar V, Churilov L, Mitchell PJ, Kleinig TJ, Yassi N, Thijs V, Wu TY, Shah DG, Ng FC, Dewey HM, Wijeratne T, Yan B, Desmond PM, Parsons MW, Donnan GA, Davis SM, Campbell BCV; EXTEND-IA TNK Investigators. Safety and Efficacy of Tenecteplase in Older Patients With Large Vessel Occlusion: A Pooled Analysis of the EXTEND-IA TNK Trials. Neurology. 2022 Mar 22;98(12):e1292-e1301. doi: 10.1212/WNL.0000000000013302. Epub 2022 Jan 11. PMID 35017305
- [Derived] Ng FC, Churilov L, Yassi N, Kleinig TJ, Thijs V, Wu T, Shah D, Dewey H, Sharma G, Desmond P, Yan B, Parsons M, Donnan G, Davis S, Mitchell P, Campbell B. Prevalence and Significance of Impaired Microvascular Tissue Reperfusion Despite Macrovascular Angiographic Reperfusion (No-Reflow). Neurology. 2022 Feb 22;98(8):e790-e801. doi: 10.1212/WNL.0000000000013210. Epub 2021 Dec 14. PMID 34906976
- [Derived] Alemseged F, Ng FC, Williams C, Puetz V, Boulouis G, Kleinig TJ, Rocco A, Wu TY, Shah D, Arba F, Kaiser D, Di Giuliano F, Morotti A, Sallustio F, Dewey HM, Bailey P, O'Brien B, Sharma G, Bush S, Dowling R, Diomedi M, Churilov L, Yan B, Parsons MW, Davis SM, Mitchell PJ, Yassi N, Campbell BCV; BATMAN study group and EXTEND IA TNK study group. Tenecteplase vs Alteplase Before Endovascular Therapy in Basilar Artery Occlusion. Neurology. 2021 Mar 2;96(9):e1272-e1277. doi: 10.1212/WNL.0000000000011520. Epub 2021 Jan 6. PMID 33408145
- [Derived] Gao L, Moodie M, Mitchell PJ, Churilov L, Kleinig TJ, Yassi N, Yan B, Parsons MW, Donnan GA, Davis SM, Campbell BCV; EXTEND-IA TNK Investigators. Cost-Effectiveness of Tenecteplase Before Thrombectomy for Ischemic Stroke. Stroke. 2020 Dec;51(12):3681-3689. doi: 10.1161/STROKEAHA.120.029666. Epub 2020 Oct 7. PMID 33023423
- [Derived] Campbell BCV, Mitchell PJ, Churilov L, Yassi N, Kleinig TJ, Dowling RJ, Yan B, Bush SJ, Dewey HM, Thijs V, Scroop R, Simpson M, Brooks M, Asadi H, Wu TY, Shah DG, Wijeratne T, Ang T, Miteff F, Levi CR, Rodrigues E, Zhao H, Salvaris P, Garcia-Esperon C, Bailey P, Rice H, de Villiers L, Brown H, Redmond K, Leggett D, Fink JN, Collecutt W, Wong AA, Muller C, Coulthard A, Mitchell K, Clouston J, Mahady K, Field D, Ma H, Phan TG, Chong W, Chandra RV, Slater LA, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Bladin CF, Sharma G, Desmond PM, Parsons MW, Donnan GA, Davis SM; EXTEND-IA TNK Investigators. Tenecteplase versus Alteplase before Thrombectomy for Ischemic Stroke. N Engl J Med. 2018 Apr 26;378(17):1573-1582. doi: 10.1056/NEJMoa1716405. PMID 29694815
- [Derived] Campbell BC, Mitchell PJ, Churilov L, Yassi N, Kleinig TJ, Yan B, Dowling RJ, Bush SJ, Dewey HM, Thijs V, Simpson M, Brooks M, Asadi H, Wu TY, Shah DG, Wijeratne T, Ang T, Miteff F, Levi C, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Bailey P, Rice H, de Villiers L, Scroop R, Collecutt W, Wong AA, Coulthard A, Barber PA, McGuinness B, Field D, Ma H, Chong W, Chandra RV, Bladin CF, Brown H, Redmond K, Leggett D, Cloud G, Madan A, Mahant N, O'Brien B, Worthington J, Parker G, Desmond PM, Parsons MW, Donnan GA, Davis SM; EXTEND-IA TNK Investigators. Tenecteplase versus alteplase before endovascular thrombectomy (EXTEND-IA TNK): A multicenter, randomized, controlled study. Int J Stroke. 2018 Apr;13(3):328-334. doi: 10.1177/1747493017733935. Epub 2017 Sep 27. PMID 28952914